CLINICAL TRIAL: NCT02652741
Title: Orodispersible Minitablets of Enalapril in Young Children With Heart Failure Due to Congenital Heart Disease
Acronym: LENA-WP09
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ethicare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-602295-02; 2015-002396-18 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure; Congenital Heart Disease
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug administration (Experimental): Enalapril Orodispersible Minitablet (ODMT), 0.25 mg or 1 mg, administered 1x/day or 2x/day for up to 8 weeks
  Interventions: Drug: Enalapril Orodispersible Minitablet

INTERVENTIONS:
Drug: Enalapril Orodispersible Minitablet — 8-weeks treatment, open, uncontrolled, PK/PD, acceptability and palatability assessments and safety assessments after Enalapril intake in form of 0.25 mg or 1 mg ODMTs
  Other Names: Enalapril ODMT

SUMMARY:
Paediatric clinical trial in 50 children, from newborn to less than 6 years of age, suffering from heart failure due to congenital heart disease, to obtain paediatric pharmacokinetic and pharmacodynamic data of enalapril and its active metabolite enalaprilat while treated for 8 weeks with enalapril in form of Orodispersible Minitablets (ODMTs), to describe the dose exposure in this patient population.

DETAILED DESCRIPTION:
This clinical trial is one of three clinical trials of the European Commission (FP7)-funded "LENA" (Labeling of Enalapril from Neonates to Adolescents) project: 50 children with heart failure due to congenital heart disease (LENA-Work Package (WP)09 Trial), and 50 children with heart failure due to dilated cardiomyopathy (LENA-WP08 Trial) get treated with an optimal dose of enalapril ODMTs for up to 8 weeks after thorough, individualised titration and get invited to join the 10 months Safety Follow-up Study (LENA-WP10 Trial).

In this WP09 Trial children from age of newborn to less than 6 years, naive to enalapril treatment or switched from an Angiotensin-Converting-Enzyme (ACE)-Inhibitor pre-treatment, receive an Initial Dose to investigate the reaction over 8 hours before a decision on the first dose level is made. Always up to 7 days later a next higher dose is given at the hospital, the patient is supervised for 4 and then always 2 hours before a decision on the prescribed dose for the next dosing period is made. In this study a target dose similar to the adult target dose (20 mg enalapril in a 70 year old adult result in 0.282 mg/kg/day enalapril) is defined. Enalapril ODMTs of 0.25 mg and 1 mg strength are available to allow for an individual dose titration scheme.

Weight-dependently, pharmacokinetic (PK) and pharmacodynamic (PD) data are collected once in a full PK/PD day over 12, respectively 6 hours, and single PK/PD samples at each Dose Titration Visit and each bi-weekly Study Control Visit until the Last Visit after 8 weeks of treatment. Blood pressure and renal monitoring is performed at each visit before deciding on the dose level for the next treatment period.

Pharmacogenomics and metabolomics exploratory studies are added as a sub-study to better understand the underlying disease, its progression as well as the impact of the ACE-inhibition on cardiac outcome and renal function.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the following Inclusion Criteria can be enrolled:

* Age from birth to less than 6 years.
* Male and female patients.
* Weight greater than 2.5 kg.
* Diagnosis of heart failure due to congenital heart disease requiring after-load reduction by drug therapy.
* Subjects may be naïve to ACE-Inhibitors.
* Subjects already on ACE-Inhibitors willing to switch to enalapril Orodispersible Minitablets.
* Patient and/or parent(s)/legal representative provided written informed consent and assent from the patient according to national legislation and as far as achievable from the child.

Exclusion Criteria:

Patients fulfilling any of the following Exclusion Criteria cannot be enrolled into this trial:

* Neonates if born < 37 weeks of gestation.
* Severe heart failure and/or end stage heart failure precluding introduction or continuation of ACE-Inhibitor.
* Too low blood pressure, e.g. ˂P5
* Uncorrected primary obstructive valvular disease, or significant systemic ventricular outflow obstruction, dilated restrictive or hypertrophic cardiomyopathy.
* Uncorrected severe peripheral stenosis of large arteries including severe coarctation of the aorta.
* Severe renal impairment with serum creatinine >2x Upper Limit of Normal (ULN) (according to the hospital's test methodology)
* History of angioedema.
* Hypersensitivity to ACE-Inhibitors.
* Concommitant medication:

  * Dual ACE-Inhibitor therapy
  * Renin inhibitors
  * Angiotensin II antagonists
  * Non-Steroidal Anti-Inflammatory Drugs (including ibuprofen) except for aspirin and paracetamol
* Already enrolled in an interventional trial with an investigational drug, unless no interference with the current study can be shown.

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Area under the Curve (AUC) of enalapril and its active metabolite enalaprilat after administration of enalapril ODMTs in children with heart failure | 0 hours to 12 hours
  Area under the Curve (AUC) of enalapril and enalaprilat are measured at first dose or at any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease (newborn to less than 6 years); descriptive pharmacokinetic investigation
Maximum Concentration (Cmax) of enalapril and its active metabolite | 0 hours to 12 hours
  Maximum Concentration (Cmax) of enalapril and enalaprilat are measured at first dose or any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease (newborn to less than 6 years); descriptive pharmacokinetic investigation
Time to Maximum Concentration (Tmax) of enalapril and its active metabolite | 0 hours to 12 hours
  Time to Maximum Concentration (Tmax) of enalapril and enalaprilat are measured at first dose or any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease (newborn to less than 6 years); descriptive pharmacokinetic investigation

SECONDARY OUTCOMES:
AUC of enalapril and its active metabolite enalaprilat after administration of enalapril ODMTs in two age-subsets of children with heart failure | 0 hours to 12 hours
  AUC of enalapril and enalaprilat are measured at first dose or any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease in the age su-sets newborn to less than 1 year and 1 to less than 6 years; descriptive pharmacokinetic investigation
Cmax of enalapril and its active metabolite enalaprilat after administration of enalapril ODMTs in two age-subsets of children with heart failure | 0 hours to 12 hours
  Cmax of enalapril and enalaprilat are measured at first dose or any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease in the age su-sets newborn to less than 1 year and 1 to less than 6 years; descriptive pharmacokinetic investigation
Tmax of enalapril and its active metabolite enalaprilat after administration of enalapril ODMTs in two age-subsets of children with heart failure | 0 hours to 12 hours
  Tmax of enalapril and enalaprilat are measured at first dose or any time during steady state to assess the bioavailability of enalapril ODMTs in young children with heart failure due to congenital heart disease in the age su-sets newborn to less than 1 year and 1 to less than 6 years; descriptive pharmacokinetic investigation
Renin | Pre-dose, 4 h post first dose, pre-dose at each Titration Visit and Study Control Visit (days 14, 28, 42) up to Last Visit (day 56)
  Renin as marker of the renin-angiotensin-aldosterone system at each study visit up to the end of treatment at 8 weeks; exploratory pharmacodynamic investigation
Angiotensin 1 | Pre-dose, 4 h post first dose, pre-dose at each Titration Visit and Study Control Visit (days 14, 28, 42) up to Last Visit (day 56)
  Angiotensin 1 as marker of the renin-angiotensin-aldosterone system at each study visit up to the end of treatment at 8 weeks; exploratory pharmacodynamic investigation
Aldosterone | Pre-dose, 4 h post first dose, pre-dose at each Titration Visit and Study Control Visit (days 14, 28, 42) up to Last Visit (day 56)
  Aldosterone as marker of the renin-angiotensin-aldosterone system at each study visit up to the end of treatment at 8 weeks; exploratory pharmacodynamic investigation
Plasma Renin Activity | Pre-dose, 4 h post first dose, pre-dose at each Titration Visit and Study Control Visit (days 14, 28, 42) up to Last Visit (day 56)
  Plasma Renin Activity as marker of the renin-angiotensin-aldosterone system at each study visit up to the end of treatment at 8 weeks; exploratory pharmacodynamic investigation
Brain natriuretic peptides (BNPs). | At Screening Visit and then pre-dose at each Titration Visit and Study Control Visit (days 14, 28, 42) up to Last Visit (day 56)
  Brain natriuretic peptides measurement as indicator of disease severity at every visit up to end of treatment at 8 weeks
Acceptability of the ODMTs | Assessment time points: at Initial Dose Visit, at one Study Control Visit (day 14, 28 or 42), at Last Visit (day 56)
  Acceptability assessment according to an age-appropriate scale
Palatability of the ODMTs | Assessment time points: at Initial Dose Visit, at one Study Control Visit (day 14, 28 or 42), at Last Visit (day 56)
  Palatability assessment according to an age-appropriate scale
Blood pressure | Pre-dose at each Visit, over 8 hours at Initial Dose Visit, over 4 hours at First Titration Visit (day 3 to 7), for 2 hours after all following Titration Visits, pre-dose at all Study Control Visits (day 14, 28, 42), at last Visit (day 56)
  Safety monitoring parameter to decide on next dose prescription level
Serum potassium | Pre-dose at each Visit: Screening Visit, Initial Dose Visit, all Titration Visits, all Study Control Visits (day 14, 28, 42) up to Last Visit (day 56)
  Renal monitoring parameter to decide on next dose prescription level
Blood urea nitrogen (BUN) | Pre-dose at each Visit: Screening Visit, Initial Dose Visit, all Titration Visits, all Study Control Visits (day 14, 28, 42) up to Last Visit (day 56)
  Renal monitoring parameter to decide on next dose prescription level
Creatinine | Pre-dose at each Visit: Screening Visit, Initial Dose Visit, all Titration Visits, all Study Control Visits (day 14, 28, 42) up to Last Visit (day 56)
  Renal monitoring parameter to decide on next dose prescription level
Micro-albuminuria | Pre-dose at each Visit: Screening Visit, Initial Dose Visit, all Titration Visits, all Study Control Visits (day 14, 28, 42) up to Last Visit (day 56)
  Renal monitoring parameter to decide on next dose prescription level
Shortening Fraction | Assessment time points: at Screening Visit and at Last Visit (day 56)
  Shortening Fraction in echocardiography
Number of patients experiencing rehospitalisation due to heart failure | During 8 weeks of treatment
  Number of patients experiencing rehospitalisation due to heart failure including the need for heart transplantation or the institution of mechanical circulatory support
Death due to worsening of the underlying disease | During 8 weeks of treatment
  Death due to worsening of the underlying disease

CONTACTS AND LOCATIONS:
Overall Officials: Milica Bajcetic, Prof,MD,PhD, Study Chair — Univerzitetska Dečja Klinika Belgrade; Ida Jovanovic, Prof,MD,PhD, Principal Investigator — Univerzitetska Dečja Klinika Belgrade; Michiel Dalinghaus, MD,PhD, Principal Investigator — Sophia Children's Hospital, Erasmus MC Rotterdam; J.M.P. J Breur, MD,PhD, Principal Investigator — Wilhelmina Children's Hospital, University Medical Center Utrecht; Christoph Male, Prof,MD,PhD, Principal Investigator — Medical University of Vienna; Michael Burch, Prof,MD,PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Trust London; András Szatmári, Prof,MD,PhD, Principal Investigator — Hungarian Paediatric Heart Centre, Göttsegen Gyorgy Hungarian Institute of Cardiology Budapest
Locations (6):
- Medical University of Vienna, Vienna, Austria
- Hungarian Paediatric Heart Centre, Göttsegen Gyorgy Hungarian Institute of Cardiology, Budapest, Hungary
- Netherlands (2):
  - Sophia Children's Hospital, Erasmus MC, Rotterdam
  - Wilhelmina Children's Hospital, University Medical Center Utrecht, Utrecht
- Univerzitetska Dečja Klinika, Belgrade, Serbia
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Serious Adverse Event information